CLINICAL TRIAL: NCT04984681
Title: Feasibility of the Mindfulness-Based Stress Reduction Intervention for Black Women Living With HIV Administrative Supplement
Brief Title: Feasibility of the Mindfulness-Based Stress Reduction Intervention for Black Women Living With HIV Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Crystal C. Lambert, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K23AT010567S; K23AT010567 (NIH)
Record Dates: First submitted 2021-07-19; First posted 2021-07-30 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections; Mild Cognitive Impairment
Keywords: HIV; Cisgender women; African American or Black; Mindfulness
MeSH Terms: conditions — HIV Infections; Cognitive Dysfunction | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Stress Reduction (Experimental): Mindfulness-based stress reduction sessions received by the treatment group will include an orientation, approximately 8 intervention sessions, and an exit interview.
  Interventions: Behavioral: Mindfulness
- Usual Care (Other): The control condition will continue receiving usual care or standard of care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Mindfulness — The traditional mindfulness intervention consists of the following: (1) orientation; (2) a series of eight weekly session of 2.5 to 3 hours; (3) a silent retreat during the between weeks 4 and 6; (4) daily home assignments including formal and informal mindfulness practices; and (5) didactic presentations on stress and the consequences of stress.
  Arms: Mindfulness-based Stress Reduction
Other: Usual Care — The control condition will continue receiving usual care or standard of care.
  Arms: Usual Care

SUMMARY:
In our Supplement Aim we will conduct a two-arm randomized pilot test of the adapted intervention compared to a usual care control group among 30 African American/Black women with HIV (15/arm) to assess the feasibility and acceptability of the mindfulness-based stress reduction among women with HIV with mild cognitive impairment. Feasibility will be assessed by our ability to (1) recruit, randomize, and retain participants and (2) deliver the intervention per the manual, as well as (3) participants adherence to home practices and assignments. Acceptability will be assessed via qualitative data (focus group input regarding participants' satisfaction with the intervention and intent to continue using the practices), as well quantitative data (satisfaction survey).

ELIGIBILITY:
Inclusion Criteria:

* Cisgender females
* HIV seropositive
* 18 years of age or older
* English speaking
* An active patient at the local HIV ambulatory clinic in Alabama.
* No history of neurological (including dementia diagnosis)
* No history of severe psychiatric (e.g., schizophrenia or bipolar disorder) disorders

Exclusion Criteria:

* Non-English speaking
* Appear temporarily impaired (e.g., intoxicated)
* Not willing to or legally unable to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We are recruiting cisgender females.
Enrollment: 30 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAB School of Nursing, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
The University of Alabama at Birmingham maintains the following universal data sharing policy for all investigators:
  1. Data will be made available, in accordance with the NIH Data Sharing Policy (http://grants.nih.gov/grants/policy/data_sharing) to all researchers in both the private and public sector free or for a nominal charge and with minimal restriction. In some cases the institution may determine that the public and the research community are better served by a licensing program whether or not patents have been filed. This may be relevant, for example, if a tool is best distributed under license to guarantee reagent availability and quality.
  2. As a means of sharing knowledge, NIH encourages grantees to arrange for publication of NIH-supported original research in primary scientific journals. We therefore will strive to publish our findings in a timely manner and acknowledge that the research was supported by the NIH.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness-based Stress Reduction | Usual Care
Started | 15 (Completed baseline assessment) | 15
Completed | 12 (Completed post-survey) | 14
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-based Stress Reduction | Usual Care | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (9.2) | 53.8 (7.4) | 55.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 15 | 30
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Mindfulness Intervention in Women With Mild Cognitive Impairment
Description: Feasibility was measured using a four-item feasibility of intervention measure. Each item is scored using a Likert-like scale ranging from "1" completely disagree to "5" completely agree. Higher scores indicate greater feasibility. The minimum total score is 4 points, and the maximum total score is 20.
Time Frame: Immediately after the intervention(which consists of an orientation followed by eight weekly sessions, consistent with MSBR interventions), the measure was collected within one week of completing the final session.
Population: This was a feasibility study. The study team was able to randomize participants. The control group did not complete the feasibility scale because they did not participate in the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Stress Reduction | Usual Care
Number analyzed (Participants) | 12 | 0
score on a scale | 18.3 (1.9) |

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Mindfulness-based Stress Reduction | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT04984681/Prot_SAP_000.pdf